CLINICAL TRIAL: NCT02547272
Title: Epidemiological Study of Intestinal Colonization With Staphylococcus Aureus in a Cohort of Adult Patients Hospitalized in Intensive Care at the University Hospital of St Etienne.
Brief Title: Epidemiological Study of Intestinal Colonization With Staphylococcus Aureus
Acronym: DigeSTAPH
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1208087; 2012-A01182-41 (Other: ANSM)
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Staphylococcus Aureus
Keywords: Intensive care; S Aureus
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — bacterial samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nasal and rectal samples: ICU patients with nasal and rectal bacterial samples for the presence of S Aureus
  Interventions: Procedure: Nasal and rectal bacterial samples

INTERVENTIONS:
Procedure: Nasal and rectal bacterial samples — Bacterial nasal and rectal samples at admission and one weekly for the presence of S Aureus

SUMMARY:
Nasal colonization with S. aureus is a risk factor for infection with this bacterium. A methodologically well conducted study of S. aureus bacteremia showed that 80% of S. aureus bacteremia with are due to the strain isolated in the nasal level. However, as part of a study coordinated by the CHU of Saint-Etienne, less than 50% of infections in prosthetic orthopedic devices have been linked to nasal carriage . Outside of exogenous infections, intestinal colonization with S. aureus could be an alternative source of endogenous infections with the waning of orthopedic surgery. In the general population, considering that about one third of the subjects were colonized with S. aureus nasal level and 1 in 5 in the intestine However the proportion of exclusive intestinal porting is not well known .

This study will analyze, among ICU patients, porting S. aureus nasal and rectal level. It will better clarify the relationship between nasal and rectal ports and the risk of developing an infection.

DETAILED DESCRIPTION:
The adult patients hospitalized in intensive care at the University Hospital of Saint-Etienne have a multiresistant bacteria porting screening at the nose and rectum at admission and then once a week. These samples will be carried unchanged way for the study but will also be a research S Aureus

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized in intensive care and benefiting from a screening multiresistant bacteria in nasal and rectal level under routine care

Exclusion Criteria:

* refusal of the patient's family

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in intensive care
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2013-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
prevalence of S. aureus colonization at rectal level | 1 month
  The presence of a colony of S. aureus on one of the samples

SECONDARY OUTCOMES:
S. aureus strains similar to nasal and rectal level | 1 month
  S. aureus strains similar in molecular typing

CONTACTS AND LOCATIONS:
Overall Officials: Philippe BERTHELOT, Md-PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No